CLINICAL TRIAL: NCT04955418
Title: Effects of Epi-no Device on Perineal Preparation and Pelvic Floor Dysfunctions
Brief Title: Effects of Epi-no Device on Pelvic Floor Dysfunctions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2.219.051
Record Dates: First submitted 2021-04-27; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Pelvic Floor Disorders; Urinary Incontinence; Dyspareunia; Lacerations Perineal
Keywords: Epi-no device; vaginal birth
MeSH Terms: conditions — Pelvic Floor Disorders; Urinary Incontinence; Dyspareunia | interventions — Physical Examination

STUDY DESIGN:
Intervention Model Description: case-control study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epi-no Group (Active Comparator): The study group was evaluated before the intervention (between 30 and 32 weeks) and 6 months after delivery.From the 34th week onwards, they performed 10 sessions (twice a week for 5 weeks) of perineal preparation with the Epi-No device. The pregnant woman was placed in the supine position and EPI-NO® was inserted into vaginal canal. After the introduction of the deflated tube, it was minimally inflated until the perception in the vaginal canal. The first 5 minutes were for perception of the pelvic floor with 10 contractions and relaxation of the perineum in order to maintain muscle strength. After 15 minutes for stretching the perineum, the device was gradually inflated and always respecting the pregnant woman's tolerance. After a total of 20 minutes, the pregnant woman was asked to relax the pelvic floor in order for the inflated device to gently exit her vaginal cavity. The perimeter was measured using a tape measure in its largest diameter.
  Interventions: Device: Epi-No®; Diagnostic Test: Evaluation
- Control Group (Placebo Comparator): The control group was evaluated only once, six month after delivery.
  Interventions: Diagnostic Test: Evaluation

INTERVENTIONS:
Device: Epi-No® — evaluation, 10 sessions (twice a week for 5 weeks) of perineal preparation with the Epi-No device and revaluation six months after delivery.
  Arms: Epi-no Group
Diagnostic Test: Evaluation — evaluation (anamnesis, childbirth data, perineometry, International Consultation on Incontinence Questionnaire - Short Form, Female Sexual Function Index) six months after vaginal delivery.

SUMMARY:
Perineal injury is the most common maternal obstetric complication associated with vaginal delivery. Perineal traumas are associated with maternal morbidity, including pain, urinary and fecal incontinence, genital prolapses, dyspareunia, physical and psychological impairment. EPI-NO is a device with the objective of preparing and training the pelvic floor for normal childbirth, this training allows smooth and slow movement along the perineal structures in the prenatal period, by causing a rapid traumatic laceration during childbirth. The objective of this study is to verify the effect of 10 pelvic stretching rows with Epi-No in preventing urinary incontinence and dyspareunia 6 months after delivery. The study group will consist of primiparous, over 18 years of age, between 30 and 32 weeks of gestation, will be evaluated before the intervention and 6 months after delivery. The control group will be evaluated only once, in the sixth month after delivery. The evaluation will consist of: anamnesis, physical examination (vaginal examination and palpation), perineometry, International Urinary Incontinence Questionnaire (ICIQ-UISF), Visual Analogue Scale for dyspareunia; Questionnaire for assessing dyspareunia Female Sexual Function Index (FSFI). Pregnant women referred for intervention will perform 10 sessions (twice a week for 5 weeks) of perineal preparation with the Epi-No device. It is expected at the end of the study to prove the effectiveness of the effect of 10 pelvic lengthening graft with Epi-No in relation to the degrees of laceration and episiotomy and, consequently, reduction of urinary incontinence and dyspareunia.

ELIGIBILITY:
Inclusion Criteria:

* primiparous
* single fetus

Exclusion Criteria:

* Patients with complaints of urinary incontinence during or before pregnancy
* hypertension and gestational diabetes
* placenta previa
* twin pregnancy
* multiparous
* patients who had undergone perineal or vaginal surgery
* patients who had urinary tract infection, genital herpes or ongoing candidiasis
* And any other diagnosis in which pregnancy becomes at risk.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Effect of birth training with Epi-no | 6 months after delivery
  Comparison the frequency of perineal tears and episiotomy between women who underwent 10 sessions of Epi-No in the pre-delivery period with women who did not undergo treatment.

SECONDARY OUTCOMES:
Pelvic floor muscle strength | 6 months after delivery
  Compare pelvic floor sensitivity and strength using perineometer between women who underwent 10 sessions of Epi-No in the pre-delivery period with women who did not undergo treatment.
Incidence of urinary incontinence and dyspareunia | 6 months after delivery
  Compare the incidence of urinary incontinence using ICIQ-SF test among women undergoing 10 sessions of pre-delivery Epi-No with women not undergoing treatment.
Incidence of dyspareunia | 6 months after delivery
  Compare the incidence of dyspareunia using FISI test among women undergoing 10 sessions of pre-delivery Epi-No with women not undergoing treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual de Londrina, Londrina, Paraná, Brazil